CLINICAL TRIAL: NCT06872983
Title: Evaluation of the Use of Synthetic Glue for Mesh Fixation in Laparoscopic Sacrocolpopexy
Acronym: LSCGlue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Samuel Tvarozek, principal investigator, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025069LSCGlue; SUp 6/25 (Other Grant/Funding Number: The University Hospital Brno Start-up grant)
Record Dates: First submitted 2025-03-03; First posted 2025-03-12 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Apical Prolapse; Sacrocolpopexy; Glue Fixation
Keywords: laparoscopic sacrocolpopexy; Tissue Adhesive; Surgical Glue; cyanoacrylate glue; implant fixation; mesh fixation
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glue mesh fixation (Experimental): The mesh will be fixed to the vaginal walls using cyanoacrylate tissue adhesive.
  Interventions: Procedure: cyanoacrylate tissue adhesive beside sutures
- Standard Care (Control): (Active Comparator): The mesh will be fixed to the vaginal walls using a standard absorbable suture.
  Interventions: Procedure: Suture

INTERVENTIONS:
Procedure: cyanoacrylate tissue adhesive beside sutures — A supracervical hysterectomy will be performed in the standard manner. Uterine amputation above the cervix will be performed with a monopolar needle or scissors. Concomitant adnexal surgery will be performed according to the presence of adnexa and the patient's request or medical indication.
  In this study group, the implant is secured to the vaginal wall with cyanoacrylate tissue adhesive. Fixation of the implant to the cervix and promontory will be identical to the control group.
  Arms: Glue mesh fixation
Procedure: Suture — A supracervical hysterectomy will be performed in the standard manner. Uterine amputation above the cervix will be performed with a monopolar needle or scissors. Concomitant adnexal surgery will be performed according to the presence of adnexa and the patient's request or medical indication. In this control group, the mesh will be fixed to the cervix with four non-absorbable sutures. In addition, the implant will be fixed to the anterior vaginal wall with four absorbable sutures and to the posterior vaginal wall with four absorbable sutures. The implant will be secured to the promontory with one non-absorbable suture.
  Arms: Standard Care (Control):

SUMMARY:
The aim of the study is to evaluate the effect of cyanoacrylate adhesive in laparoscopic sacrocolpopexy, which is the gold standard treatment for apical prolapse. The procedure is predominantly performed using minimally invasive techniques, such as laparoscopic or robotic methods. However, the operative time for this procedure often exceeds 180 minutes due to its technical complexity. Although the experience level of the surgical team can lead to a decrease in operative time, there is a concerning increase in the risk of postoperative complications as the duration of surgery extends. One strategy to mitigate overall operative time is to reduce the fixation time of the implant to the vaginal wall.

Standard fixation involves using several sutures, but alternative fixation methods, including barbed sutures and cyanoacrylate adhesives, may demonstrate a reduction in fixation time. While there are only a few studies available on the use of cyanoacrylate adhesives for implant fixation, they generally indicate that this method is safe and can achieve an objective success rate of over 96% in resolving apical descent. However, the reported operative time using glue varies significantly across studies, ranging from 69 to 173 minutes.

The aim of the current study is to assess the impact of a synthetic cyanoacrylate-based tissue adhesive on various factors, including implant fixation time, overall length of surgery, short- and long-term postoperative complications, risk of prolapse recurrence, and the cost-effectiveness of this method in comparison to traditional laparoscopic sutures. This will be conducted as a randomized prospective monocentric study that includes patients aged 18 to 75 years diagnosed with pelvic organ descent grade 2 or higher. Notably, individuals requiring uterine preservation, having undergone previous hysterectomy, or with precancerous or malignant uterine diseases will be excluded.

The surgical approach will involve fixing the implant to the vaginal wall with cyanoacrylate adhesive in the target group, along with non-absorbable sutures. In contrast, the control group will follow traditional fixation methods using absorbable sutures in addition to non-absorbable ones. The study will evaluate outcomes using various questionnaires, including the POPQ for anatomical effect and PFDI-20 for subjective discomfort, while also assessing postoperative pain through the VAS scale.

Expected results include a targeted reduction in implant fixation time by at least 20 minutes and a comprehensive evaluation of the method's cost-effectiveness based on reports from Brno University Hospital. This study is significant as it represents the first prospective randomized trial to investigate the effects of cyanoacrylate adhesive on operative time and cost-effectiveness compared to conventional suturing in laparoscopic sacrocolpopexy

ELIGIBILITY:
Inclusion Criteria:

* Sufficient knowledge of the Czech language
* Pelvic organs prolapse of second stage or higher according to POPQ classification (POPQ ≥ 2)
* Patients indicated for laparoscopic sacropexy - sacrocervicopexy with concomitant supracervical hysterectomy

Exclusion Criteria:

* Patients requesting uterine preservation
* Patients with previous hysterectomy
* Patients with premalignancy or malignancy of the female reproductive organs
* Concomitant urethropexy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender females
Enrollment: 40 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The duration of fixation of the implant to the walls of the vagina with the adhesive in comparison to the standard suture. | Enrollment to surgery: 4-8 weeks
  To determine whether or not the duration of fixation of the implant to the anterior and posterior vaginal walls using adhesive is statistically significantly shorter in minutes compared to standard fixation using sutures. The statistical evaluation will be based on time measured with a stopwatch (minutes). The time is measured from the start of fixation of the implant to the vaginal walls until it is completely anchored to the vaginal walls. This objective does not evaluate the time required for complete fixation of the implant including fixation to the promotorium, but only the time required to fix the implant to the vagina.

SECONDARY OUTCOMES:
Total mesh fixation time | Enrollment to surgery: 4-8 weeks
  The total time (in minutes) required to manipulate the implant - from its insertion into the abdominal cavity to its fixation to the promontory (including fixation to the cervix and vaginal walls). The total time required for implant fixation between the two groups will be analyzed.
Total time of the operation | Enrollment to surgery: 4-8 weeks
  The total operative time (in minutes) is defined as the interval from the initial placement of all laparoscopic trocars to their subsequent removal. A statistical evaluation will be conducted to compare the total time required to complete the surgical procedure between the two groups.
Peri- and post-operative complications | From surgery to 12 months
  All perioperative and all postoperative complications will be monitored. The severity of postoperative complications will be assessed according to the Clavien-Dindo classification.
Perioperative pain intensity and analgetic utilization | intervals: 6, 24 and 48 hours after surgery
  All patients will receive analgesics during the postoperative period in accordance with the prevailing therapeutic protocol at the Gynecology and Obstetrics Clinic of the University Hospital Brno. The intensity of pain experienced by patients in the postoperative period will be documented using the Visual Analogue Scale (VAS 0-10) at 6, 24, and 48 hours following surgery. Furthermore, the necessity for opioid analgesics to manage pain will be documented. Subsequent analyses will compare the two groups with respect to the necessity of analgesic and opioid analgesic utilization in the early postoperative period.
Recurrence rate of pelvic organ prolapse | 6 to 12 months
  In the late postoperative period (6 and 12 months), the recurrence of pelvic organ prolapse will be assessed in each compartment using a standardized Pelvic Organ Prolapse Quantification System (POP-Q). A finding of Ba ≥ -1, Bp ≥ -1, or C > TVL/2 is considered a recurrence. A statistical comparison will be conducted to evaluate the incidence of recurrence between the two groups.
The degree of bother and distress caused by pelvic floor symptoms. | change from baseline to 8-12 weeks, 6 and 12 months
  Pelvic Floor Disability Index (PFDI-20) - This is a short form that provides a comprehensive assessment of the impact of pelvic floor disorders on women's quality of life. The PFDI-20 consists of 3 scales, including the Urinary Distress Inventory-6 (UDI-6), the Pelvic Organ Prolapse Distress Inventory-6 (POPDI-6) and the Colorectal-Anal Distress Inventory-8 (CRADI-8). The PFDI-20 serves the role of both a symptom inventory and a measure of the degree of bother and distress caused by the broad array of pelvic floor symptoms. Lower scores indicate less distress caused by the presence of pelvic floor dysfunction symptoms. A comparative analysis of the groups will be performed in relation to the change in subjective perception of difficulties, as assessed by the PFDI-20, after surgery at predetermined intervals.
The impact of a floor dysfunction on the quality of life | change from baseline to 8-12 weeks, 6 and 12 months
  The Pelvic Floor Impact Questionnaire-7 (PFIQ-7) is a health-related quality-of-life questionnaire to assess life impact in women with pelvic floor disorders. The questionnaire incorporates scales from the Urinary Impact Questionnaire (UIQ-7), the Pelvic Organ Prolapse Impact Questionnaire (POPIQ-7) and the Colorectal-Anal Impact Questionnaire-7 (CRAIQ-7). The emphasis of the questionnaire is directed towards the impact of pelvic discomfort on the day-to-day activities of the individual. The PFIQ-7 is a valuable tool for measuring changes in symptom severity over time, both before and after treatment, and as such is a useful addition to the existing array of health-related quality-of-life questionnaires. A comparative analysis of the groups will be performed in relation to the change in health-related quality of life, as assessed by the PFIQ-7, after surgery at predetermined intervals.
Quality of life of women with urinary incontinence | change from baseline to 8-12 weeks, 6 and 12 months
  International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) - A questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women. where higher scores indicate greater symptom severity. This tool determines the change from baseline - improvement or deterioration of urinary incontinence and will be used as a screening tool for de-novo urinary incontinence after surgery. Additionally, it includes a self-diagnostic item to help identify the type of incontinence. A comparative analysis of the groups will be performed in relation to urinary incontinence and de-novo urinary incontinence after surgery at predetermined intervals.
Sexual function evaluation | change from baseline to 8-12 weeks, 6 and 12 months
  The PISQ-IR (Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, IUGA-Revised) is a validated evaluation tool for the assessment of female sexual function in women with female pelvic floor disorders. The PISQ-IR is composed of multiple domains that address different aspects of sexual function. The single summary score will be used to evaluate change from baseline in both groups. Moreover, the individual domains of the questionnaire will be evaluated separately. A comparative analysis of the groups will be performed in relation to the change in sexual functions after surgery.
The patient's subjective impression of improvement since surgery | change from baseline to 8-12 weeks, 6 and 12 months
  The Patient Global Imression of Improvement (PGI-I) is a global index that may be used to rate the response of a condition to a therapy. The PGI-I indicates overall satisfaction with post-operative condition based on this scale:
  1. Very much better; 2. Much better; 3. A little better; 4. No change; 5. A little worse; 6. Much worse; 7. Very much worse.
  The PGI-I will be utilized to evaluate patient satisfaction with the postoperative status in comparison to the preoperative status. The patient will complete the PGI-I at predefined postoperative intervals 8-12 weeks, 6 and 12 months. Subsequently, a comparative analysis of the two groups will be performed on patient satisfaction with the postoperative condition.
Position of the implant | change from baseline to 8-12 weeks, 6 and 12 months
  The position of the implant will be measured using transperineal and transvaginal ultrasound. The position will be measured as a distance (in millimeters) of the lowermost visible mesh echogenicity from the bladder neck on the anterior vaginal wall and from the perineum on the posterior vaginal wall. A comparative analysis of the implant position in the two study groups will be conducted to ascertain whether the method of fixation exerts an influence on implant placement.
Mesh related complications | From surgery to 12 months
  Any postoperative mesh complications associated with the implant will be recorded using a Prosthesis/Graft Complication Classification Code for both groups. The calculation will be made using the official IUGA/ICS classification tool available from: https://www.ics.org/complication
Total cost of care using adhesive fixation versus standard laparoscopic intracorporeal suturing | 3 months after surgery
  This part of the study aims to evaluate the total cost of care using adhesive fixation versus standard laparoscopic intracorporeal suturing. The cost of adhesive materials and applicators is significant compared to suture-only methods; however, if adhesive use reduces operative time considerably, financial savings may be achieved. The Controlling Department of University Hospital Brno will provide reports to assess total hospitalization costs, expressed in Czech crowns, which include material, operating room, and postoperative care expenses. These reports will be available three months post-discharge. The study seeks to compare hospitalization costs for adhesive fixation and conventional procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Tvarozek, MD, Principal Investigator — Department of Obstetrics and Gynecology, University Hospital Brno, Brno, Czech Republic
Locations (1):
- Brno University Hospital, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR